CLINICAL TRIAL: NCT06799715
Title: Assessments of Metabolic Responses to Acute Oral Administration of Sucrose, Glucose, and Fructose in Healthy Humans
Brief Title: Assessments of Metabolic Responses to Acute Oral Administration of Sucrose, Glucose, and Fructose
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SuGluFru
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Gastrointestinal Hormones; Glycemic Control; Blood Coagulation Function; Gastric Emptying
MeSH Terms: interventions — Sucrose; Glucose; Fructose; Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sucrose (Active Comparator): 20 volunteers receive 33.5g sucrose dissolved in 300mL water as a drink.
  Interventions: Dietary Supplement: Sucrose
- Glucose (Active Comparator): 20 volunteers receive 33.5g glucose dissolved in 300mL water as a drink.
  Interventions: Dietary Supplement: Glucose
- Fructose (Active Comparator): 20 volunteers receive 33.5g fructose dissolved in 300mL water as a drink.
  Interventions: Dietary Supplement: Fructose
- Water (Placebo Comparator): 20 volunteers receive 300mL water as a drink.
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Sucrose — 33.5g sucrose dissolved in 300mL tap water
  Other Names: Saccharose
  Arms: Sucrose
Dietary Supplement: Glucose — 33.5g glucose dissolved in 300mL tap water
  Other Names: Dextrose
  Arms: Glucose
Dietary Supplement: Fructose — 33.5g fructose dissolved in 300mL tap water
  Arms: Fructose
Dietary Supplement: Water — 300mL water
  Arms: Water

SUMMARY:
This project aims to compare the acute metabolic effects of the three sweeteners sucrose, glucose, and fructose on GI hormones (GLP-1, PYY, CCK, and ghrelin).

Furthermore, glycemic control, erythritol and xylitol concentrations, blood coagulation function , blood lipids, uric acid, high-sensitive C-reactive protein (hsCRP), complete blood count, gastric emptying, appetite-related sensations, and GI symptoms will be investigated.

DETAILED DESCRIPTION:
Sugar should not be defined by origin (added sugar, free sugar, simple sugar) but rather by chemical structure (sucrose, glucose, fructose, etc.). Although the disaccharide sucrose is hydrolysed by sucrase into its monosaccharides glucose and fructose, the administration of each of the three sweeteners alone results in different metabolic effects.

Although sucrose, glucose, and fructose are long known sweeteners in food and beverages and their metabolic effects have been extensively studied, there are still no comprehensive studies comparing the three sweeteners in a whole range of parameters. The main inconsistency in the literature is the study design which influences the outcomes. It is important to differentiate whether it is an acute or chronic study, whether the participants are adults or children, are healthy or have T2DM, have normal weight, overweight or obesity, whether the dosage is chosen to be isocaloric or isosweet, whether there is a control group or whether the sweeteners are administered orally or intragastrical.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, non-diabetic (glycated hemoglobin (HbA1c) < 5.7%, fasting glucose < 5.6 mmol/L), and normal weight participants with a body-mass index (BMI) of 19.0-24.9 kg/m2, parameters of complete blood count within normal range
* Age 18-55 years
* Stable body weight (± 5%) for at least three months
* Able to give informed consent as documented by signature

Exclusion Criteria:

* Fructose intolerance
* Any pre-existing diet (e.g., vegetarian diet, vegan diet, sugar free diet, paleo diet, Atkins diet, ketogenic diet) that deviates from normal eating habits
* Regular consumption (>1/ week) of erythritol or xylitol
* Regular intake of medications, except contraceptives
* Pre-existing impairment of blood coagulation/thrombocyte function (e.g. hereditary, regular intake of anti-coagulant agents (e.g. NSAIDs, heparin, warfarin, etc.))Chronic or clinically relevant acute infections/diseases
* Substance abuse (more than 1 glass wine/beer per day; regular consumption of cannabis, consumption of cocaine, heroin, etc.), regular smoking
* Pregnancy: although no contraindication, pregnancy might influence metabolic state. Women who are pregnant or have the intention to become pregnant during the course of the study are excluded. In female participants a urine pregnancy test is carried out upon screening.
* Shift worker
* Participation in another study with investigational drug within the 30 days preceding and during the present study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Effect of sucrose, glucose, fructose, and water on the GI hormone response - GLP-1 | Blood will be drawn at the following timepoints: : -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration)
  Plasma GLP-1 will be measured with a commercially available immunoassay kit (MILLIPLEX® MAP; Millipore Corporation, Billerica, MA, USA).
Effect of sucrose, glucose, fructose, and water on the GI hormone response - PYY | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  PYY-3-36 will be quantified using a non-radioactive high sensitive sandwich ELISA (Millipore - # EZHPYYT66K).
Effect of sucrose, glucose, fructose, and water on the GI hormone response - CCK | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Plasma cholecystokinin (CCK) levels will be measured with a sensitive radioimmunoassay using a highly specific antiserum (No. 92128)
Effect of sucrose, glucose, fructose, and water on the GI hormone response - Ghrelin | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Octanoylated ghrelin will be measured by a radioimmunoassay with 125I [Tyr24] human ghrelin as tracer and a rabbit antibody against human ghrelin (final dilution 1/100000), which does not cross-react with desoctanoylated ghrelin.

SECONDARY OUTCOMES:
Effects on glycemic control - plasma glucose | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Glucose will be measured by a glucose oxidase method (Rothen Medizinische Laboratorien AG, Basel, Switzerland).
Effects on glycemic control - plasma insulin | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Insulin will be quantified using a chemiluminescent microparticle immunoassay (chemiflex) reagent kit (#8k41; Abbott) and the relative light units detected by the ARCHITECT optical system (model: CI4100; Abbott).
Effects on glycemic control - plasma c-peptide | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  C-peptide will be measured with a commercially available sandwich ELISA kit from Millipore (Millipore - # EZHCP-20K).
Effects on glycemic control - plasma glucagon | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Glucagon concentrations in plasma will be measured after extraction of plasma with 70% ethanol (vol/vol, final concentration). The antibody is directed against the C-terminus of the glucagon molecule (antibody code no. 4305) and therefore mainly measures glucagon of pancreatic origin.
Effects on erythritol concentrations | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Erythritol concentrations will be measured by GC-MS/MS (Gas Chromatography Tandem Mass Spectrometry).
Effects on xylitol concentrations | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 120, and 180minutes (after administration).
  Xylitol concentrations will be measured by GC-MS/MS (Gas Chromatography Tandem Mass Spectrometry).
Effects on blood coagulation function - p-selectin | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180 minutes (after administration).
  Plasma concentrations of p-selectin will be measured using a commercially available ELISA-kit.
Effects on blood coagulation function - sVCAM1 | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180 minutes (after administration).
  Plasma concentrations ofsVCAM1 will be measured using a commercially available ELISA-kit.
Effects on blood coagulation function - PF-4 | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180 minutes (after administration).
  Plasma concentrations of PF-4 will be measured using a commercially available ELISA-kit.
Effects on blood coagulation function - D-Dimers | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180 minutes (after administration).
  D-Dimers will be measured using an antigen-test.
Effects on blood lipids | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120 and 180 minutes (after administration).
  Analyses of blood lipids are carried out in the hospital laboratory.
Effects on uric acid | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180 minutes (after administration).
  Analyses of uric acid are carried out in the hospital laboratory.
Effects on hsCRP | Blood will be drawn at the following time points: -10 and -1 minutes (before administration) and 30, 60, 90, 120, and 180minutes (after administration).
  Concentrations of hsCRP will be measured by Rothen Laboratory in Basel.
Effects on gastric emptying rate | Breath samples will be drawn at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 240minutes (after administration).
  Gastric emptying rate will be determined using a 13C-sodium acetate breath test.
Effects on appetite-related sensations | Visual analogue scales will be recorded at the following time points: -10 and -1 minutes (before administration) and 15, 30, 45, 60, 90, 105, 120, and 180 minutes (after administration).
  Appetite perceptions (feelings of: a) hunger, b) satiety) are assessed by visual analogue scale (VAS). Visual analogue scales consist of a horizontal, unstructured, 10-cm line representing the minimum (0.0 points) to the maximum rating (10.0 points). Subjects assign a vertical mark across the line to indicate the magnitude of their subjective sensation at the present time point. The measurement is quantified by the distance from the left end of the line (minimum rating) to the subject's vertical mark.
Effects on GI tolerance | GI tolerance will be recorded atthe following time points: -10 minutes (before administration) and 30, 60, 90,120, 180, and 240 minutes (after administration).
  GI symptoms will be assessed by use of a checklist including the following questions: abdominal pain, nausea, vomiting, diarrhoea, borborygmi, abdominal distension, eructation and increased flatus.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Christin Meyer-Gerspach, PD, PhD, Principal Investigator — St. Clara Research Ltd.
Locations (1):
- St. Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No